CLINICAL TRIAL: NCT00421187
Title: Phase III Study of 3 Sequential Doses (10 mg/kg, 5 mg/kg, and 5 mg/kg) vs 3 mg/kg/Day of AmBisome® in the Management of Culture-negative Neutropenic Fever Unresponsive to Antibiotics
Brief Title: Ambisome and Management of Culture-negative Neutropenic Fever Unresponsive to Antibiotics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit subjects in the Turkey site.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Lazaros Poughias, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-MM-131-0162
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2008-04

CONDITIONS: Febrile Neutropenia
Keywords: Antibiotic resistant neutropenic fever; ARNF; Ambisome; Liposomal amphotericin B
MeSH Terms: conditions — Febrile Neutropenia | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AmBisome® will be given on day 0 (10 mg/kg), day 2 (5 mg/kg), and day 5 (5 mg/kg)
  Interventions: Drug: Liposomal amphotericin B (AmBisome®)
- 2 (Active Comparator): AmBisome as a constant daily dose of 3 mg/kg for a maximum of 14 days or until the resolution of fever and neutropenia
  Interventions: Drug: Liposomal amphotericin B (AmBisome®)

INTERVENTIONS:
Drug: Liposomal amphotericin B (AmBisome®)
  Arms: 1
Drug: Liposomal amphotericin B (AmBisome®)
  Other Names: Ambisome
  Arms: 2

SUMMARY:
Administration of a single high dose (10 mg/kg) of AmBisome® no later than 72 hours after ARNF onset followed by two 5 mg/kg doses on days 2 and 5 may provide sustained tissue levels of amphotericin B that are as mycologically effective as those provided after administering the standard daily dose of 3 mg/kg/day. The new dosing regimen is anticipated to be equally clinically effective compared with the standard AmBisome® regimen when given for the duration of neutropenic fever in patients with ARNF. In addition, the degree and incidence of nephrotoxicity are predicted to be lower with the 3 sequential dose regimen compared to daily dosing with 3 mg/kg because of the lower cumulative dosage (20 mg/kg versus 42 mg/kg, respectively), which is 1 contributing factor for the development of acute renal failure. Furthermore, the lower cumulative dose may be a cost-effective strategy for the treatment of patients with ARNF.

DETAILED DESCRIPTION:
This is a phase III, multicenter, randomized, open-label study. One center in the United Arab Emirates and 1 center in Turkey will participate in this trial and approximately 50 patients will be recruited.

Patients will be adults with hematological malignancies undergoing chemotherapy for leukemia or lymphoma. These patients will be treated with AmBisome® until resolution of fever and neutropenia or for a maximum of 14 days.

Patients will be randomized to receive AmBisome 10 mg/kg on treatment day 0 followed by 5 mg/kg on days 2 and 5 or AmBisome 3 mg/kg/day for 14 days. Study medication will be administered during the period of ARNF until resolution of fever and neutropenia and/or a minimum of 14 days. At the end of the 14-day trial period, each patient will be classified as having responded or not responded to the treatment according to the criteria for response given below.

Patients will be examined daily for evidence of drug toxicity or intolerance and for the development of an IFI. Vital signs will be recorded every 6 hours if the patient is stable or more frequently if there is evidence of clinical deterioration. In the event of a clinical IFI (i.e., development of a halo sign or positive fungal blood cultures), the patient will be withdrawn from the study, classified as treatment failure, and receive antifungal treatment with either caspofungin or voriconazole. Daily clinical observations will ensure rapid detection of such an event in accordance with standard IDSA guidelines4. Patients who show clinical deterioration (i.e., increasing dyspnea, hypotension) but exhibit no definite evidence of an IFI may also be classified as treatment failures. Patients with evidence of biochemical and/or clinical drug toxicity will be withdrawn from the study and appropriate management will be given.

For patients who remain febrile after 14 days but who are otherwise stable and have no discernable cause for the fever, continuation of treatment with AmBisome 3 mg/kg/day or treatment with another antifungal drug treatment, antibiotic, or discontinuation of antimicrobial therapy will be undertaken at the discretion of the investigator. Patients who meet these criteria will have a thorough diagnostic evaluation to investigate the cause of their fever.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study. Adult patients with hematologic malignancy undergoing chemotherapy for leukemia or lymphoma will be recruited into this study from 2 centers provided the following inclusion criteria are fulfilled:

  * Male or female
  * Age ≥ 18 years
  * Neutropenia (< 0.5 x 109 cells/L)
  * Received empiric antibiotic treatment for 3 days for blood culture negative infection
  * Persistent fever of ≥ 38°C
  * No known IFI at baseline during this neutropenic episode. However, patients with "missed" evidence of IFI (features absent at randomization but evidence within 48 hours [eg, positive chest computerized tomography (CT)]) will complete the randomized treatment and kinetic measurements
  * No antifungal prophylaxis or treatment in this hospital admission or for the past 30 days
  * Baseline liver function tests ≤ 10 times the upper limit of normal and baseline creatinine ≤ 2 times the upper limit of normal
  * No known hypersensitivity to amphotericin B or LAMB or any of its constituents, in particular known history of anaphylactic reaction to amphotericin B or LAMB or any of its constituents
  * Females of childbearing potential (less than 2 years post menopausal) must be surgically incapable of pregnancy, or practicing an acceptable method of birth control with a negative pregnancy test (blood or urine) at baseline
  * Ability to comply with all study requirements
  * Written informed consent

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

  * Evidence of proven, probably or possible invasive fungal infection
  * Chronic invasive fungal infection, defined as signs/symptoms of invasive fungal infection present for >4 weeks preceding entry into study
  * Prior systemic therapy greater or equal to 4 days with any polyene anti-fungal agent within 30 days of study enrollment
  * Prior systemic therapy with non-polyenes (i.e., azole or echinochandin derivatives) for the current ARNF. (Prior systemic anti-fungal therapy with non-polyene derivatives for prophylaxis or as empiric therapy for febrile neutropenia is permissible.)
  * Use of another investigational, unlicensed drug within 30 days of screening or concurrent participation in another clinical trial using an investigational, unlicensed drug.
  * Serum creatinine > 2x upper limit of normal (ULN)
  * Serum ALT or AST > 5x ULN
  * History of allergy or serious adverse reaction to any polyene anti-fungal agent.
  * Patients who have a positive blood culture within 5 days before day 0 with a clinically significant organism isolated from the peripheral blood, who despite appropriate antibiotics have persistent positive cultures
  * Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
PK Profile of the dosing regimen under study (AUC, Cmax, Cmin, and etc.) | throughout

SECONDARY OUTCOMES:
Proportion of patients with defervescence (temperature < 38°C for ≥ 48 hours) occurring during neutropenia | throughout
Time to defervescence from start of study entry and from time fever first recorded | throughout
Proportion of patients with emergence of an IFI during AmBisome® treatment | throughout
Survival during hospital admission | throughout
Survival at 14 days after study initiation | Day 14
Proportion of patients with treatment-emergent adverse events | throughout
Proportion of patients with treatment-emergent adverse events related to study drug | throughout
Proportion of patients with post-baseline toxicity grading changes in each laboratory test (those graded according to the protocol). | throughout

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros Poughias, MD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Athens, Greece